CLINICAL TRIAL: NCT00005363
Title: Ambulatory Blood Pressure and Prognosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4250; R01HL048945 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To continue a prospective study of the ability of ambulatory blood pressure to predict cardiovascular morbidity in patients with mild hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

This was a continuation of a prospective study of the ability of ambulatory blood pressure to predict cardiovascular morbidity in patients with mild hypertension, which was first started in 1978.

DESIGN NARRATIVE:

Predictor variables evaluated at entry to the longitudinal study included clinic and ambulatory blood pressures (including measures of pressure level and variability in different settings), left ventricular mass index (LVMI, determined by echocardiography), renin-sodium profile, and other cardiovascular risk factors (e.g., cholesterol and smoking). During follow-up, blood pressure, treatment status, BMI, and clinical course were evaluated. Outcome measures were definite cardiovascular morbid events, defined as sudden cardiac death, myocardial infarction, stroke, congestive heart failure, and coronary artery revascularization. The main hypotheses tested were that ambulatory blood pressure would give a better prediction of outcome than clinic pressure, and that patients with white coat hypertension (defined as a high clinic pressure and normal ambulatory pressure) would be at low risk relative to patients with sustained hypertension. Initial results in 729 patients initially studied between 1978 and 1985 using Cox survival analysis showed that the four most significant predictors of morbid events were daytime blood pressure variability, age, male sex, and serum cholesterol. Patients with white coat hypertension appeared to be at a level of risk intermediate between normotensives and sustained hypertensives, but the differences were not yet significant. Expansion of the cohort size to include patients evaluated initially between 1985 and 1990 provided nearly 2,000 patients altogether, which together with the longer follow-up of the initial cohort provided a sufficient number of morbid events to identify the predictive significance of the different blood pressure measures, and their interaction with other risk factors.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-08; Study Completion 1994-07 (Actual)

REFERENCES:
- [Background] Loupal G. [Gastrolithiasis in a llama]. Berl Munch Tierarztl Wochenschr. 1982 Jan 1;95(1):14-6. No abstract available. German. PMID 7059338
- [Background] James GD, Toledano T, Datz G, Pickering TG. Factors influencing the awake-sleep difference in ambulatory blood pressure: main effects and sex differences. J Hum Hypertens. 1995 Oct;9(10):821-6. PMID 8576898
- [Background] Devereux RB, de Simone G, Ganau A, Roman MJ. Left ventricular hypertrophy and geometric remodeling in hypertension: stimuli, functional consequences and prognostic implications. J Hypertens Suppl. 1994 Dec;12(10):S117-27. PMID 7769482
- [Background] Devereux RB, Roman MJ, Ganau A, de Simone G, Okin PM, Kligfield P. Cardiac and arterial hypertrophy and atherosclerosis in hypertension. Hypertension. 1994 Jun;23(6 Pt 1):802-9. doi: 10.1161/01.hyp.23.6.802. PMID 8206580
- [Background] Devereux RB, James GD, Pickering TG. What is normal blood pressure? Comparison of ambulatory pressure level and variability in patients with normal or abnormal left ventricular geometry. Am J Hypertens. 1993 Jun;6(6 Pt 2):211S-215S. PMID 8347321
- [Background] Pickering TG, James GD. Determinants and consequences of the diurnal rhythm of blood pressure. Am J Hypertens. 1993 Jun;6(6 Pt 2):166S-169S. doi: 10.1093/ajh/6.6.166s. PMID 8347311
- [Background] Devereux RB. Left ventricular geometry, pathophysiology and prognosis. J Am Coll Cardiol. 1995 Mar 15;25(4):885-7. doi: 10.1016/0735-1097(94)00547-4. No abstract available. PMID 7884092
- [Background] Pickering TG, James GD. Ambulatory blood pressure and prognosis. J Hypertens Suppl. 1994 Nov;12(8):S29-33. PMID 7707152